CLINICAL TRIAL: NCT03901599
Title: Feasibility of Protective Ventilation Based on the Alveolar Ventilation in Paediatric Anaesthesiology and Intensive Care.
Brief Title: Protective Ventilation Based on Alveolar Ventilation in Children
Acronym: PROVENTIPED
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0114
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia; Peroperative Complication
MeSH Terms: conditions — Intraoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Children between 5-10Kg: Children with a body weight between 5-10Kg
  Interventions: Other: Alveolar ventilation monitoring estimated by the capnographic ventilation
- Children between 10-20Kg: Children with a body weight between 10-20Kg
  Interventions: Other: Alveolar ventilation monitoring estimated by the capnographic ventilation
- Children between 20-40Kg: Children with a body weight between 20-40Kg
  Interventions: Other: Alveolar ventilation monitoring estimated by the capnographic ventilation

INTERVENTIONS:
Other: Alveolar ventilation monitoring estimated by the capnographic ventilation — Children are monitored using end-tidal CO2, Transcutaneous CO2 and volumetric capnographic. Respiratory rate is set using textbooks and guidelines (pediatric advanced life support). The physician in charge adapts the volume to target a CO2 between 38 and 42 mmHg. Data are recorded after a stabilization period of at least 5 minutes.

SUMMARY:
Protective ventilation decreased morbidity and mortality in adults' patients and is now a standard of care in intensive care unit and in anesthesiology. In children, there is no evidence in the literature to recommend protective ventilation during anaesthesia. Moreover the ratio of instrumental dead space to tidal volume is higher in children than in adults. Therefore, it is difficult to propose an "optimal" tidal volume for all children. The objective of this study is to evaluate the use of alveolar ventilation (estimated by the volumetric capnography) in children under anesthesia. The hypothesis is that in children, alveolar ventilation reported to ideal body weight is a constant to maintain normocarbia, unlike the tidal volume.

ELIGIBILITY:
Inclusion Criteria:

* Children aged < 12 and
* Weight between 5 and 40kg
* General anesthesia
* Non-opposition of parents or legal guardians

Exclusion Criteria:

* History of bronchodysplasia or laryngo tracheo malacia, cyanotic heart disease or neuromuscular disease
* Airleaks > 10%
* Bronchospasm during anesthesia

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2019-10-27 (Actual); Study Completion 2019-10-27 (Actual)

PRIMARY OUTCOMES:
Determination of target alveolar minute volume to maintain normocapnia in children without mechanical ventilation. | 5 minutes after hemodynamic and ventilatory stabilization period
  The minute alveolar ventilation estimated by the volumetric capnography reported to the ideal body weight based on 100 breaths (expressed in ml/Kg/min).

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric anesthesia division, Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gardon A, De Queiroz Siqueira M, Cerceuil E, Bouhamri N, Chassard D, Baudin F. Alveolar target ventilation and dead space in children under anaesthesia: The proventiped cohort study. Eur J Anaesthesiol. 2023 Jul 1;40(7):495-500. doi: 10.1097/EJA.0000000000001832. Epub 2023 Apr 12. PMID 37052073